CLINICAL TRIAL: NCT03259477
Title: Renal Functional Reserve Change of Precise Segmental Versus Complete Renal Arterial Clamping During Laparoscopic Partial Nephrectomy for Clinical T1 Renal Cell Carcinoma
Brief Title: RFR Change of Precise Segmental Versus Complete Renal Arterial Clamping During LPN for Clinical T1 RCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, ou tongwen, chairman of urology, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: otw-20170804-02
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Renal Cell Carcinoma
Keywords: laparoscopic partial nephrectomy; precise segmental renal arterial clamping; renal cell carcinoma; renal functional reserve
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: Some participants with clinical T1 renal cell carcinoma(RCC) undergo precise segmental during laparoscopic partial nephrectomy and the others undergo complete renal arterial clamping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- precise segmental clamping (Experimental): These participants with clinical T1 renal cell carcinoma(RCC) undergo precise segmental renal arterial clamping during laparoscopic partial nephrectomy.
  Interventions: Procedure: precise segmental renal arterial clamping; Procedure: laparoscopic partial nephrectomy
- complete clamping (Active Comparator): These participants with clinical T1 renal cell carcinoma(RCC) undergo complete renal arterial clamping during laparoscopic partial nephrectomy.
  Interventions: Procedure: laparoscopic partial nephrectomy

INTERVENTIONS:
Procedure: precise segmental renal arterial clamping — Precise segmental renal artery clamping eliminates global renal ischemia by performing highly selective clamping of single or multiple segmental arteries.
  Arms: precise segmental clamping
Procedure: laparoscopic partial nephrectomy — Laparoscopic partial nephrectomy (LPN) has been widely adopted as a minimally invasive nephron-sparing surgery for clinical T1 renal cell carcinoma(RCC).

SUMMARY:
Renal functional reserve may be better in patients with clinical T1 renal cell carcinoma(RCC) undergoing laparoscopic partial nephrectomy with precise segmental renal artery clamping than those with complete renal arterial clamping.

DETAILED DESCRIPTION:
Renal functional reserve (RFR) describes the capacity of the intact nephron mass to increase glomerular filtration rate(GFR) from baseline in response to stimuli (e.g., protein load).We hypothesized that renal functional reserve may be better in patients with clinical T1 renal cell carcinoma(RCC) undergoing laparoscopic partial(LPN) nephrectomy with precise segmental renal artery clamping than those with complete renal arterial clamping.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥18 2.Estimated GFR >30 mL/min/1.73m2 3.Anticipated intraoperative warm ischemic time ≤30 min 4.Subjects who signed informed consent forms

Exclusion Criteria:

1. Allergy to iothalamate, shellfish or iodine
2. Use of metformin or amiodarone
3. intraoperative warm ischemic time >30 min
4. Inability to maintain a stable regimen of medications which affect GFR for > one week prior to participation (e.g. non-steroidal anti-inflammatory drugs, angiotensin converting enzyme inhibitors, angiotensin receptor blockers)
5. Use of medications which directly affect elimination of creatinine (e.g. cimetidine and trimethoprim)
6. Acute exacerbation of asthma or chronic obstructive pulmonary disease within 3 months requiring hospitalization or oral steroid therapy
7. Inadequate intravenous access
8. Severe anemia (Hct <21%)
9. Acute kidney injury (rise in creatinine to ≥1.5 times the previous baseline or by ≥ 0.3 mg/dL on most recent labs prior to enrollment)
10. History of contrast-induced nephropathy
11. Hyperthyroidism
12. Pheochromocytoma
13. Sickle cell disease
14. Urinary retention or incontinence
15. Status post organ transplant
16. Pregnancy or active breast feeding
17. Cognitive impairment with inability to give consent
18. Institutionalized status

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Renal Functional Reserve change | 3 month after surgery.
  Change in renal functional reserve after laparoscopic partial nephrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Tongwen Ou, MD., Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, China